CLINICAL TRIAL: NCT00673868
Title: A Phase I-II Randomized Trial to Examine the Clinical, Immunologic and Virologic Effects of CMV Specific CTL When Used for Prophylaxis Against CMV Disease in Recipients of Allogeneic, T Cell Depleted Stem Cell Transplants
Brief Title: Cytomegalovirus (CMV) Specific Cytotoxic T Lymphocytes (CTL) When Used for Prophylaxis Against CMV in Recipients of Allogeneic, T Cell Depleted Stem Cell Transplants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Milton S. Hershey Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 26769
Record Dates: First submitted 2008-05-01; First posted 2008-05-07 (Estimated); Last update posted 2017-07-02 (Actual); Status verified 2017-06

CONDITIONS: Cytomegalovirus Infections
MeSH Terms: conditions — Cytomegalovirus Infections

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental)
  Interventions: Biological: CMV Specific Cytotoxic T Lymphocytes
- 2 (No Intervention)

INTERVENTIONS:
Biological: CMV Specific Cytotoxic T Lymphocytes — CMV Specific Cytotoxic T Lymphocytes will be infused between days 30 and 40 post-transplant at a dose ranging from 2- 5 x e5 cells/kg.
  Arms: 1

SUMMARY:
This study examines the immunologic and virologic effects of prophylactic CMV specific CTL in recipients of T cell depleted stem cell transplant (TCD SCT) at Duke University Medical Center (DUMC), by measuring levels of CMV DNA and virus specific T cell precursors at intervals post-infusion.

DETAILED DESCRIPTION:
Human cytomegalovirus (CMV) is a benign infectious agent in the normal host, but in immunocompromised individuals, such as recipients of stem cell or organ transplants, this virus is a major cause of morbidity and mortality. While pharmacologic agents exist to treat CMV disease, these medications have numerous side effects, the most serious of which is myelosuppression. Considering the risk associated with persistent infection and the potential for CMV specific CTL to restore immunity, we propose to study the immunologic and virologic effects of CMV pp65 specific CTL given to SCT recipients prophylactically, levels of CMV pp65 specific CTL and CMV DNA will be measured from CTL recipients and a control group randomized to not receive CTL.

All treatments will be given at Duke University Medical Center (DUMC).

1. Patients will have a complete set of vital signs and physical examination prior to each infusion. Pulse oximetry will be monitored prior to, during, and for 30 minutes after the T-cell infusion. Thirty minutes prior to the CTL infusion, patients will be pre-medicated with 15 mg/kg (maximum 1 g) of acetaminophen p.o. and 1.0 mg/kg diphenhydramine I.V. (maximum 50 mg). Cells will be thawed in the Cell Therapy lab at DUMC, an aliquot sent for gram stain and culture, and viability will be determined. Cells with > 70 % viability will be transferred to the clinical unit and infused over 5-10 minutes.
2. CMV CTL will be infused when available between days 30 and 40 post-transplant at a dose ranging from 2- 5 x 105 cells/kg. This dose range was established since there may be variability in the numbers of CTL expanded from these donors.

This trial intended to be a Phase 1/2 trial, but it never progressed to Phase 2 before completion.

ELIGIBILITY:
Inclusion Criteria:

* Any allogeneic stem cell transplant recipient > 2 years of age who is CMV sero-positive and has a CMV sero-positive donor,
* Bilirubin < 2.0 mg/dl; SGOT/SGPT < 2.5 X normal.
* Creatinine clearance > 50 cc/min as estimated by patient's serum creatinine, weight, and age.
* Pulse oximetry > 95% on no supplemental oxygen.
* ECOG performance status < 2; for patients, 16 years of age, Lansky performance status >70%.

Exclusion Criteria:

* Sero-negative patients with a history of GVHD of grade II or greater by the Glucksberg crireria (protocol Appendix I) at or prior to day +30 of current stem cell transplant are excluded.
* Patients who have received a prior stem cell transplant are excluded.
* Patients who are moribund or who because of cardiac, pulmonary, renal, hepatic or neurologic dysfunction are not expected to survive one month.
* Subjects receiving systemic immunosuppressive agents for the treatment of GVHD at the time of the CTL infusion will be excluded from receiving CTL, and subjects randomized to not receive CTL will also be removed from study if at the time of the CTL infusion they require systemic immunosuppression for treatment of GVHD
* Donors must be negative for HIV-1, HIV-2, and HTLV-2, and have passed all screening tests for hepatitis.

Ages: 2 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2007-10; Primary Completion 2008-08-06 (Actual); Study Completion 2008-08-06 (Actual)

PRIMARY OUTCOMES:
The primary objective is to characterize CMV specific immunity in subjects receiving and in those randomized to not receive CMV CTL. We will characterize CMV CTLp frequencies and bulk cytotoxicity at days 30 and 60 post infusion. | one year

SECONDARY OUTCOMES:
To characterize the time to develop CMV specific immunity in pts. receiving and not receiving CTL by assessing CMV CTL | one year
To determine the CMV epitopes recognized by donors | one year
To characterize the levels of CMV DNA in recipients of CMV CTL and non CTL | one year

CONTACTS AND LOCATIONS:
Overall Officials: Kenneth G. Lucas, MD, Principal Investigator — Penn State University
Locations (1):
- Penn State University, Hershey, Pennsylvania, United States